CLINICAL TRIAL: NCT00118261
Title: A Phase IB Study in Patients With Metastatic Colorectal Cancer to Evaluate Pharmacodynamic Effects of Erlotinib and Safety and Efficacy of Erlotinib in Combination With Modified FOLFOX6 (mFOLFOX6) and Bevacizumab
Brief Title: Erlotinib, Modified FOLFOX6, and Bevacizumab as First-Line Therapy Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Smitha Krishnamurthi, Principal Investigator, Case Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2204; P30CA043703 (NIH); CASE2204 (Other: Case Comprehensive Cancer Center); NCI-2009-01287 (Other: NCI/CTRP)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Cancer
Keywords: stage IV rectal cancer; stage IV colon cancer; recurrent rectal cancer; recurrent colon cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms; Colonic Neoplasms | interventions — Bevacizumab; Erlotinib Hydrochloride; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib, modified FOLFOX6, and bevacizumab (Experimental)
  Interventions: Biological: bevacizumab; Drug: erlotinib hydrochloride; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin

INTERVENTIONS:
Biological: bevacizumab — Beginning in course 3, patients also receive bevacizumab IV over 30 minutes. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Drug: erlotinib hydrochloride — Courses 1-3: oral erlotinib once daily on days 1-14. Patients who do not develop grade 2 toxicity after the first 3 courses (6 weeks) will have their erlotinib dose escalated. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Drug: fluorouracil — Starting with course 2: fluorouracil IV continuously over 46 hours on days 1 and 2. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Drug: leucovorin calcium — Starting with course 2: Leucovorin calcium IV over 2 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Drug: oxaliplatin — Starting with course 2: oxaliplatin IV over 2 hours on day 1. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Erlotinib may help chemotherapy work better by making tumor cells more sensitive to the drugs. Giving erlotinib together with combination chemotherapy and bevacizumab may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of erlotinib when given together with combination chemotherapy and bevacizumab as first-line therapy in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of erlotinib, mFOLFOX6, and bevacizumab in patients with metastatic colorectal cancer.
* Determine the efficacy of this regimen in these patients.
* Determine the feasibility of escalating the dose of erlotinib in order to maximize the likelihood of developing a grade 2 skin rash in select patients.

OUTLINE: This is a multicenter study.

* Single-agent erlotinib: Patients receive oral erlotinib once daily on days 1-14 (course 1).
* Erlotinib, modified FOLFOX6, and bevacizumab chemotherapy: Patients receive oral erlotinib* once daily on days 1-14, oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1, and fluorouracil IV continuously over 46 hours on days 1 and 2 in course 2. Beginning in course 3, patients also receive bevacizumab IV over 30 minutes. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.

NOTE: Patients who do not develop grade 2 toxicity after the first 3 courses (6 weeks) will have their erlotinib dose escalated.

PROJECTED ACCRUAL: A total of 22 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed colorectal cancer

  * Biopsy-accessible metastatic disease
* Measurable disease
* No CNS metastases

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* WBC ≥ 4,000/mm^3 OR
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 10 g/dL
* No bleeding disorder

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* Albumin ≥ 2.5 g/dL

Renal

* Creatinine ≤ 1.5 mg/dL
* Urine protein:creatine ratio < 1.0

Cardiovascular

* Blood pressure ≤ 150/100 mmHg
* No arterial thrombotic event within the past 6 months
* No New York Heart Association grade II-IV congestive heart failure

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 1 month after completion of study treatment
* No other malignancy within the past 3 years except nonmelanoma skin cancer, carcinoma in situ of the cervix, or other malignancy with < 10% chance of relapse within 3 years
* No uncontrolled infection
* No severe uncontrolled illness that would preclude study participation
* No peripheral neuropathy interfering with function
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No serious non-healing wound, ulcer, or bone fracture

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No concurrent sargramostim (GM-CSF)

Chemotherapy

* No prior chemotherapy, including oxaliplatin, for metastatic disease
* Prior adjuvant oxaliplatin allowed provided disease progressed > 12 months after completion of oxaliplatin
* At least 3 weeks since prior cytotoxic chemotherapy (6 weeks for mitomycin or nitrosoureas)

  * No more than 2 courses of prior mitomycin
* No concurrent chemotherapy

Endocrine therapy

* No concurrent anticancer hormonal therapy

Radiotherapy

* At least 2 weeks since prior radiotherapy
* No prior radiotherapy to > 15% of bone marrow
* No concurrent radiotherapy

Surgery

* At least 4 weeks since prior major surgery
* At least 1 week since prior minor surgery

Other

* Recovered from prior therapy
* No prior epidermal growth factor receptor inhibitor therapy
* No other concurrent antineoplastic or antitumor therapy
* No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2005-03; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Number of patients that develop study drug related toxicity | 3 courses (6 weeks)
  Dose-limiting toxicities will be tracked in the first three cycles. The occurrence of DLT in 2 of the first 6 patients, 3 of the first 9 patients, or 4 of the first 12 patients (whichever occurs soonest)will require that subsequent patients are enrolled to the study at 100 mg erlotinib daily.

SECONDARY OUTCOMES:
Patient Response to Treatment Measured by RECIST Criteria | 3 courses (6 weeks)
  The overall response is the number of participants who experience a confirmed complete (CR) or partial response (PR) of the total analysis population. Per the Response Evaluation Criteria In Solid Tumors (RECIST): CR = all detectable tumor has disappeared, PR = a >=30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum, Progressive disease (PD) = a >=20% increase in target lesions, Stable Disease = small changes that do not meet previously given criteria.
Number of patients that can increase the erlotinib dose to 200mg | 14 days
  The number of patients requiring an increase in erlotinib dose to 200 mg will be reported as well as the toxicities observed at 200 mg daily erlotinib, the median onset to grade 2 or higher rash and diarrhea at 200 mg erlotinib, and the number of patients requiring a decrease in erlotinib from 200 mg.

CONTACTS AND LOCATIONS:
Overall Officials: Smitha Krishnamurthi, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - MetroHealth Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - UHHS Chagrin Highlands Medical Center, Cleveland, Ohio